CLINICAL TRIAL: NCT06596083
Title: The Effects of Ketone Ester Supplementation During a 5 Week Live High, Train Low Altitude Training Camp
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Chiel Poffé, postdoctoral researcher, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: S67562
Record Dates: First submitted 2024-08-27; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hypoxia; Exogenous Ketosis
Keywords: Altitude training camp; Exercise; Live high, train low; EPO
MeSH Terms: conditions — Hypoxia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will go through the entire 5 week training camp and 1 week follow up while taking either ketone ester supplements (KE) or an isocaloric placebo (CON).
Who Masked: Participant, Investigator
Masking Description: Participants and investigators are blinded from the experimental condition (KE or CON). Supplements are provided in non transparent tubes and the control supplement is identical in taste and viscosity to the ketone supplement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Comparator (Placebo Comparator): Training intervention: 5 weeks of live high, train low followed by an additional 1 week of reduced training (to simulate preparation for an upcoming event or race) Dietary intervention: placebo supplement
  Interventions: Dietary Supplement: Placebo supplement
- Experimental group (Experimental): Training intervention: 5 weeks of live high, train low followed by an additional 1 week of reduced training (to simulate preparation for an upcoming event or race) Dietary intervention: Ketone ester supplement
  Interventions: Dietary Supplement: Ketone ester supplement

INTERVENTIONS:
Dietary Supplement: Placebo supplement — oral supplement containing: 16.4 grams of medium chained triglycerides, 1mM or sucrose octaacetate and water
  Arms: Placebo Comparator
Dietary Supplement: Ketone ester supplement — Oral supplement containing: 25 grams of pure (R)-3-hydroxybutyl-(R)-3-hydroxybutyrate ketone monoester drink
  Arms: Experimental group

SUMMARY:
This study aims to investigate the effects of post-exercise and pre-sleep exogenous ketosis via oral ketone ester supplementation during a 5 week simulated altitude training camp.

DETAILED DESCRIPTION:
Altitude training camps, where you train at sea level but live at altitude, have become a popular way for athletes to prepare for upcoming races or events. The main aim of such training camps is to benefit from the adaptations following prolonged hypoxic exposure (increased EPO concentrations leading to an increase in oxygen carrying capacity in the blood). Recently, ketone bodies have been shown to cause similar adaptations. Therefore, this study aims to investigate whether the combination of exogenous ketosis and an altitude training camp is more beneficial compared to an altitude training camp on its own.

Participants will follow a 5 week simulated altitude training camp where they spend 75 hours per week at altitude (2000-3000 meters), while taking ketone or placebo supplements after every training sessions and before going to sleep. During these 5 weeks, they will adhere to a prescribed training plan, consisting of 5 to 7 training sessions per week. Before, after and 1 week after the training camp, their exercise performance, EPO concentrations, hemoglobin mass and VO2max will be tested.

ELIGIBILITY:
Inclusion Criteria:

* Physically fit and regularly involved in physical activity (2-5h per week)
* Good health status confirmed by a medical screening
* Non-smoking

Exclusion Criteria:

* Any kind of injury/pathology that is a contra-indication to perform high-intensity exercise
* Any kind of injury/pathology that is a contra-indication for exposure to hypoxia
* Ongoing pregnancy or breastfeeding
* intake of any medication or nutritional supplement that is proven to affect exercise performance during the last month prior to the start of the study
* Involvement in elite athletic training at a semi-professional or professional level
* Exposure to altitudes higher than 1500 m during the 3 months prior to the start of the study
* Blood ferritin levels below 30 ng/mL
* Current participation in another research trial
* Any other argument to believe that the subject is unlikely to succesfully complete the full study protocol

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-09-10 (Estimated); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Total hemoglobin mass | Day 0, Day 35, Day 42
  Using the optimized CO-re-breathing method, total hemoglobin mass will be estimated
Skeletal muscle capillarization | Day 0, Day 35, Day 42
  Changes in muscle capillarization are measured using immunohistochemical anlyses
Cycling exercise performance | Day 0, Day 35, Day 42
  maximal average power output during a 30 minute time trial, cycling efficiency test and repeated sprint test

SECONDARY OUTCOMES:
Maximal oxygen uptake (VO2max) | Day 0, Day 35, Day 42
  Using ergospirometry VO2max will be measured during a graded exercise test
Change in peripheral blood flow | Day 0, Day 35, Day 42
  Measured using duplex ultrasonography
Serum EPO concentrations | Day 0, day1, week1, week2, week3, week4, week5, day35, day42
  Serum EPO concentrations will be measured using a commercially available ELISA kit
Sleep Architecture | Day 0, day1, week 3, day35, day42
  Polysomnography will be used to measure sleep architecture

CONTACTS AND LOCATIONS:
Overall Officials: Chiel Poffé, Principal Investigator — KU Leuven
Locations (1):
- KU Leuven, Leuven, Vlaams-Brabant, Belgium